CLINICAL TRIAL: NCT07298902
Title: Non-Invasive Deep Brain Neuromodulation for Smoking Cessation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Xiaoming Du, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-25-1070
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Nicotine Addiction
Keywords: low intensity focused ultrasound
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active low intensity focused ultrasound (LIFU) (Experimental): Participants in this group will receive active LIFU treatment
  Interventions: Device: Low intensity focused ultrasound with active stimulations
- Sham LIFU (Sham Comparator): Participants in this group will receive sham LIFU treatment
  Interventions: Device: low intensity focused ultrasound with sham stimulations

INTERVENTIONS:
Device: Low intensity focused ultrasound with active stimulations — Participants will receive two LIFU sessions a week for 4 weeks.
  Arms: Active low intensity focused ultrasound (LIFU)
Device: low intensity focused ultrasound with sham stimulations — Participants will receive two LIFU sessions a week for 4 weeks.
  Arms: Sham LIFU

SUMMARY:
This study will develop novel low intensity focused ultrasound (LIFU) therapy to help people to quit cigarette smoking. Smoking is associated with cancers of the lung. Available smoking cessation methods help many to quit. However, for the many who continue to smoke despite the strong desire to quit and after exhausting existing therapeutic approaches, new treatment methods are needed. Without more effective treatment, many will continue to smoke, and our progress on cancer prevention through smoking cessation may decelerate as these associated cancer risks will remain. Brain imaging research has identified specific areas of the brain linked to severe nicotine addiction, but up to now there are no effective ways to directly target most of these deeper brain regions. LIFU is a new and safe method to modulate brain functions that can either inhibit overactive activity or restore normal activity levels. The purpose of this study is to provide a novel ultrasound-based neuromodulation strategy for smoking cessation in people who have difficulty to quit smoking despite numerous serious attempts in their lives. LIFU works by sending acoustic pressure modulating neural activity in the human brain.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a smoker for 5 or more years and within 20 to 60 years of age
2. Must not meet exclusion criteria for MRI scanning (e.g., non-fixed magnetizable objects)
3. Must not have ongoing unstable medical, neurological or psychiatric illness as determined by a combination of history, medical record, and/or examination.
4. Must be a current smoker with average of 5 cigarettes or more a day for the last month or longer.
5. Report 3 or more trials of smoking cessation attempts using nicotine replacement, e-cig, TMS, varenicline or other smoking cessation drugs, psychotherapy or other means.

Exclusion Criteria:

1. Failed TMS screening questionnaire.
2. Significant alcohol or other drug use (substance dependence within the recent months) or positive urine toxicology screen for substance not prescribed other than nicotine or marijuana dependence.
3. Cannot refrain from using alcohol and/or marijuana 24 hours or more prior to experiments.
4. Taking > 400 mg clozapine/day and not on anti-seizure medication(s) with sufficient dose.
5. Woman who is pregnant (child-bearing potential but not on contraceptive and missing menstrual period; or by self-report; or by positive pregnancy test) or has had unprotected sexual intercourse without birth control in the last 4 weeks.
6. In ongoing smoking cessation treatment, clinical trial, or nicotine replacements (except for the current study)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Cigarette per day (CPD) | Baseline, session 1 (about 1-2 days after baseline), session 8 (about 4 weeks after baseline), and 1-week follow up (about 5 weeks after baseline).
  Cigarette per day (CPD) is measured to index smoking reduction and cessation.
Brain connectivity as indicated by resting state functional connectivity (rsFC) value as assessed by functional magnetic resonance imaging (fMRI) | session 1 (about 1-2 days after baseline) and session 8 (about 4 weeks after baseline).
  The strength of rsFC from fMRI is used to represent the brain activities that are corresponding to the transcranial magnetic stimulation (TMS) effect on smoking reduction/cessation.

SECONDARY OUTCOMES:
End-expired carbon monoxide (CO) | Baseline, session 1 (about 1-2 days after baseline), session 8 (about 4 weeks after baseline), and 1-week follow up (about 5 weeks after baseline).
  End-expired CO measure is an instant measure of smoking status, with higher CO level indicating more severe recent smoking behavior.
Urinary cotinine level | Baseline, session 1 (about 1-2 days after baseline), session 8 (about 4 weeks after baseline), and 1-week follow up (about 5 weeks after baseline).
  Urinary cotinine is an index of smoking status, with higher cotinine concentrations indicating more severe smoking behavior.
Quit rate (%) | Session 1 (about 1-2 days after baseline), session 8 (about 4 weeks after baseline), and 1-week follow up (about 5 weeks after baseline).
  Quit rate is an index of smoking cessation effects of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Du, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No